CLINICAL TRIAL: NCT02613533
Title: What is the Effect of the "Water Drinking Test" on Patients With Narrow Angles on the Day of Their Scheduled Laser Iridotomy?
Brief Title: Water Drinking Test in Patients With Occludable Angle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jonathon Myers, Principle Investigator, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-988E
Record Dates: First submitted 2015-08-10; First posted 2015-11-24 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Narrow Angle Glaucoma Study Group (Experimental): Subjects will be given 10ml/kg of water over 15 min prior to surgery and Intra-ocular pressure measurement (IOP) is checked every 15 min before and after surgical procedure.
  Interventions: Other: Intra-ocular pressure measurement (IOP)

INTERVENTIONS:
Other: Intra-ocular pressure measurement (IOP) — Subjects will be given 10ml/kg of water over 15 min prior to laser peripheral iridotomy (LPI) surgery and Intra-ocular pressure (IOP) is tested every 15 min before and after surgical procedure

SUMMARY:
The water drinking test (WDT), is a predictive test that has been used to detect primary open angle glaucoma and recently has been demonstrated as a predictor of the diurnal tension curve. Clinically accurate provocative tests for asymptomatic eyes with shallow anterior chambers and narrow angles are highly desirable to detect patients prone to angle closure glaucoma. The aim of this pilot study is to evaluate the possible role of water drinking test in patients with narrow angles who are scheduled for prophylactic laser iridotomy.

DETAILED DESCRIPTION:
This prospective case series will investigate the effects of the WDT on subjects with narrow anterior chamber angles on the day of their scheduled laser iridotomy. The angle configuration and IOP will be monitored following the WDT. Twenty patients with occludable angles will be enrolled in this study. After measuring the baseline IOP, weight and height, the patients will be asked to drink 10ml/kg water over 15 minutes (equal to approximately 0.33 ounces of water for every 2.2 pounds of weight or 2 ½ cups for a 150 lb. individual) and their IOP will be checked every 15 minutes up to one hour after drinking the water. This will be repeated after performing a laser iridotomy. The data obtained, mainly IOP and gonioscopic findings, will be analyzed using statistical tests and compared to historical controls of the WDT without narrow angles, and laser iridotomy subjects without the WDT.

ELIGIBILITY:
Inclusion Criteria:

* narrow angle judged to be at risk of attack by the treating physician, with one or more quadrants not open to the sclera spur on gonioscopy
* age between 21 and 90 years
* ability to give informed consent.

Exclusion Criteria:

* baseline IOP higher than 21 mm Hg with or without medication
* other causes of glaucoma, such as pseudoexfoliative and pigmentary glaucomas
* previous treatment with argon laser or selective laser trabeculoplasty
* previous refractive sugary; (5) pregnant women; (6) congestive heart failure
* renal failure or urinary retention issues; (8) corneal abnormalities preventing reliable IOP measurement
* non-glaucomatous optic neuropathy
* prior refractive surgery or other issues preventing accurate Goldmann applanation tonometry
* prior intraocular surgery

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Intra-ocular pressure measurement | every 15 minutes before and after surgery for upto an hour
  Twenty patients with occludable angles will be enrolled in this study. After measuring the baseline Intra-ocular pressure, weight and height, the patients will be asked to drink 10ml/kg water over 15 minutes (equal to approximately 2 ½ cups for a 150 lb. individual) and their intra-ocular pressure (IOP) will be checked every 15 minutes up to one hour after drinking the water. This will be repeated after performing a laser peripheral iridotomy (LPI). The data obtained, mainly Intra-ocular pressure will be analyzed using statistical tests and compared to historical controls of the WDT without narrow angles, and laser iridotomy subjects without the WDT.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Myers, MD, Principal Investigator — Wills Eye
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
A manuscript has been accepted for publication in Patient Preference and Adherence.